CLINICAL TRIAL: NCT03299374
Title: Estudio Comparativo de Los Beneficios Del Método Pilates Frente a un Programa específico de prevención de caídas
Brief Title: Effectiveness of the Pilates Method to Prevent and Reduce Falls in Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Jose María Blasco Igual, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pilates _FB
Record Dates: First submitted 2017-09-26; First posted 2017-10-03 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Aging Problems
Keywords: Pilates; Balance; Falls; Older people

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are informed, so masking is not ensured Outcomes evaluator masked Physiotherapist none masked External adviser masked (randomization and data analysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Falls Group (Active Comparator): Falls prevention intervention
  Interventions: Other: Fall prevention intervention
- Pilates Group (Experimental): Pilates intervention
  Interventions: Other: Pilates Intervention

INTERVENTIONS:
Other: Pilates Intervention — Intervention based on Pilates principles
  Arms: Pilates Group
Other: Fall prevention intervention — Intervention based on principles to prevent falls
  Arms: Falls Group

SUMMARY:
The present research aims at evidencing the effect of one of the training methodologies increasingly demanded by the older adult, and used to promote, maintain and enhance physical and biopsychosocial aspects. Consequently, we intend to base the evidence supporting Pilates as an effective method in the following specific aspects: balance, prevention and reduction of falls, and improvement of the quality of life in the older adult

ELIGIBILITY:
Inclusion Criteria:

* Subjects +60 years.
* Subjects without cognitive impairment that prevent from performing interventions. A score in the Mini-Cognitive Examination of Lobo has to be equal or greater than 20 points.
* Subjects without physical impairment that prevent from performing interventions, or can directly influence the evaluation of the balance abilities (i.e., vestibular pathologies, amputated limbs, etc.)
* Subjects willing to participate, and have read, understood and signed an informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Falls calendar | 1 year follow-up
  Number of falls

SECONDARY OUTCOMES:
Falls Efficacy Scale International | change from baseline to end of intervention (4 month) and follow-up (1 year)
  Risk of falls
Timed UP and Go Test | change from baseline to end of intervention (4 month) and follow-up (1 year)
  Dynamic balance
Functional Reach Test | change from baseline to end of intervention (4 month) and follow-up (1 year)
  Stability
One Leg stance | change from baseline to end of intervention (4 month) and follow-up (1 year)
  Static Balance
Euro Quality of Life 5 Dimension | change from baseline to end of intervention (4 month) and follow-up (1 year)
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Blasco, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain